CLINICAL TRIAL: NCT06547268
Title: Heart@Home: Advancing the Science of Pediatric Interstage Home Monitoring
Brief Title: Advancing the Science of Pediatric Interstage Home Monitoring
Acronym: Heart@Home
Status: Terminated | Type: Observational
Why Stopped: Changes to sensor to test
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Sibel Health Inc. (Industry)
Responsible Party: Principal Investigator, Carolyn Foster, Assistant Professor of Pediatrics, Northwestern University
Other Study IDs: 2023-6397
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Heart Defects, Congenital
Keywords: Heart Defects, Congenital; Digital Health
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Home monitoring program patients: Patients enrolled in the study are those patients who are already enrolled in (or are being discharged with) home monitoring in an existing program
  Interventions: Device: Wireless sensor and platform

INTERVENTIONS:
Device: Wireless sensor and platform — Skin-mounted sensor that pairs with tablet platform
  Other Names: Arc

SUMMARY:
The overall goal of this study is to understand the feasibility of using a wireless sensor device (instead of a wired device) to collect information used to monitor children with heart conditions at home.

DETAILED DESCRIPTION:
The goal of this study is to examine how well continuous sensor-based monitoring performs at detecting physiologic data in infants with single ventricle physiology at home compared to existing approaches, in manner that is feasible and acceptable to patients' families. Performance features of interest include how the data compares to family measurements, whether it correlates with parents' observable symptoms, and how this approach may be integrated into home life and health system workflows. The investigators will also explore whether the collected data can be used to develop predictive analytics for acute deterioration and/or advanced chronic cardiopulmonary management compared to what is currently being done in remote patient monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Receiving active remote patient monitoring (RPM) in Lurie's Tele-Interstage Home Monitoring Program.
* Age 0-2 years of age at enrollment.
* In the opinion of the investigator, parent or legally authorized guardian, and participant, the participant and (when relevant) family can follow study procedures.

Exclusion Criteria:

* Is going to discontinue RPM before their enrollment would end (i.e., within 14 days).
* Skin breakdown or severe rash at the site of sensor placement.
* Patient without a parental guardian to consent.
* The patient is in active hospice or similar end-of-life care.
* The patient will be living in a long-term institution or transitional facility.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children receiving remote patient monitoring in tele-interstage home monitoring program.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Physiologic measurements | up to 14 days per patient of data collection
  Physiologic data waveform morphology

SECONDARY OUTCOMES:
Systems Usability Score | up to 14 days per patient of data collection
  Score from 0 (min) to 100 (max) of usability with higher is better (100=perfect).
Utilization | up to 14 days per patient of data collection
  Emergency departnment use

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn C Foster, MD, MS, Principal Investigator — Ann and Robert H. Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Data requests will be reviewed by PI if the occur.

REFERENCES:
- [Background] Foster C, Schinasi D, Kan K, Macy M, Wheeler D, Curfman A. Remote Monitoring of Patient- and Family-Generated Health Data in Pediatrics. Pediatrics. 2022 Feb 1;149(2):e2021054137. doi: 10.1542/peds.2021-054137. PMID 35102417
- [Background] Foster CC, Steltzer M, Snyder A, Alden C, Helner K, Schinasi DA, Bohling K, Allen K. Integrated Multimodality Telemedicine to Enhance In-Home Care of Infants During the Interstage Period. Pediatr Cardiol. 2021 Feb;42(2):349-360. doi: 10.1007/s00246-020-02489-7. Epub 2020 Oct 20. PMID 33079264
- [Background] Rudd NA, Ghanayem NS, Hill GD, Lambert LM, Mussatto KA, Nieves JA, Robinson S, Shirali G, Steltzer MM, Uzark K, Pike NA; American Heart Association Council on Cardiovascular and Stroke Nursing; Council on Lifelong Congenital Heart Disease and Heart Health in the Young; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Clinical Cardiology; and Council on Lifestyle and Cardiometabolic Health. Interstage Home Monitoring for Infants With Single Ventricle Heart Disease: Education and Management: A Scientific Statement From the American Heart Association. J Am Heart Assoc. 2020 Aug 18;9(16):e014548. doi: 10.1161/JAHA.119.014548. Epub 2020 Aug 11. PMID 32777961